CLINICAL TRIAL: NCT02891967
Title: One-year Clinical Evaluation of Bulk-fill Resin Composite Using FDI Criteria in Comparison to Conventional Incremental Posterior Restoration
Brief Title: One-year Clinical Evaluation of Bulk-fill Versus Conventional Incremental Posterior Restoration by FDI Criteria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mary Sabry Tawfik Tadros, researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CEBD-CU-08-184
Record Dates: First submitted 2016-08-30; First posted 2016-09-08 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Post Dental Restoration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bulk full composite (3M) (Other): bulk fill composite in posterior class one cavities
  Interventions: Other: bulk fill composite; Other: Nano resin composite (K Z350 xt)
- Incremental packing composite resin (Other): Nano resin composite (K Z350 xt) restoration in class one cavities
  Interventions: Other: bulk fill composite; Other: Nano resin composite (K Z350 xt)

INTERVENTIONS:
Other: bulk fill composite — cavities will be incrementally layered with resin composite and each increment will be cured as directed by the manufacturer with the light curing unit (XL 3000; 3M/eSPe), with an energy higher than 450 mW/cm² (±50 mw/cm²)
Other: Nano resin composite (K Z350 xt) — cavities will be restored by bulk fill composite (3M ESPE) as one increment then will be cured as directed by the manufacturer with the light curing unit.

SUMMARY:
restoring posterior teeth by bulk fll and nanofill composite and clinical evaluation of performance and durability of both restorations during one year follow up

DETAILED DESCRIPTION:
The treated cavities will be divided into 2 groups, cavities will be incrementally layered with resin composite and each increment will be cured as directed by the manufacturer with the light curing unit (XL 3000; 3M/eSPe), with an energy higher than 450 mW/cm² (±50 mw/cm²) and other group of cavities will be restored by bulk fill composite (3M ESPE) as one increment then will be cured as directed by the manufacturer with the light curing unit.

Articulation will be checked carefully with an articulating paper and occlusal adjustments will be performed using flame shaped carbide and diamond finishing burs (DENTSPLY) using water spray, restorations will be finished occlusally with finishing burs and finally polished with aluminium oxide polishing paste and a rubber cup (DENTSPLY).

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene.Patients must show no signs of orofacial pain. The presence of molar teeth requiring composite restorations for the treatment of primary carious lesions

Exclusion Criteria:

* Teeth with abnormal periapical anatomy or caries that will be likely to result in very deep restorations. Teeth with old restorations or severely destructed dental crowns.Tempro-mandibular joint problems involving symptomatic pain.Pregnancy or breast feeding, acute and chronic systemic diseases, immune-compromised patients

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-03 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
clinical performance and durability of restoration | one year
  Outcome measure is Clinical performance and durability of composite resin restoration, Device for measurement is FDI criteria , Unit of measurement is Ranking system has 5 scores for each different criterion. Either restoration is clinically excellent, or good, or sufficient, or unsatisfactory, or clinically poor.

CONTACTS AND LOCATIONS:
Overall Officials: Mary ST Tadros, Phd, Study Chair — Cairo University
Locations (1):
- Mary, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No